CLINICAL TRIAL: NCT03210454
Title: Evaluation Of The Effect Of Marketing Interventions For Women On Economic Empowerment And Risk Of Intimate Partner Violence In Colombia
Brief Title: Evaluation of Marketing Interventions in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kathryn Yount, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00083606
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Gender Based Violence; Intimate Partner Violence
MeSH Terms: interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Intervention Model Description: The randomization occurs at the farmer's association level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group 1 (Experimental): Farmers associations, including men and women, will be randomized to receive the smallholder marketing intervention.
  Interventions: Other: Smallholder Marketing
- Treatment Group 2 (Experimental): Farmers associations, including men and women, will be randomized to receive the smallholder marketing intervention combined with the intimate partner violence (IPV) prevention training.
  Interventions: Other: Smallholder Marketing; Other: Intimate Partner Violence (IPV) Prevention Training
- Comparison Group 3 (No Intervention): Women involved with farmers's associations that work independently of World Food Programmes (WFP's) assistance.

INTERVENTIONS:
Other: Smallholder Marketing — The smallholder marketing intervention involves product purchasing (e.g., bananas, beans, goats, eggs) from smallholder farmers' associations through WFP's large procurement procedures. WFP is will also provide technical training on topics such as sustainable farming practices, quality control, and business practices.
  Arms: Treatment Group 1; Treatment Group 2
Other: Intimate Partner Violence (IPV) Prevention Training — IPV prevention training involves 24 hours of gender training (gender equality and rights, economic empowerment, gender-based violence prevention), and 8 hours of nutrition and food security training (with a focus on gender).
  Arms: Treatment Group 2

SUMMARY:
The proposed project seeks to implement a cluster-randomized controlled trial (RCT) to measure the impact of increasing women´s incomes and providing gender equality trainings on women´s empowerment and risk of intimate partner violence (IPV) in Colombia. This project will be the first in Latin America to evaluate rigorously the impact of a marketing intervention, alone and combined with IPV prevention training. The knowledge generated from this evaluation has the potential to identify the most effective solutions to empower women, as well as to drive transformative change in current approaches to reduce IPV and promote gender equality in highly vulnerable populations in Colombia, and worldwide.

DETAILED DESCRIPTION:
The proposed project seeks to implement a cluster-randomized controlled trial (RCT) to measure the impact of increasing women´s incomes and providing gender equality trainings on women´s empowerment and risk of intimate partner violence (IPV) in Colombia. This project will be the first in Latin America to evaluate rigorously the impact of a marketing intervention, alone and combined with IPV prevention training. The knowledge generated from this evaluation has the potential to identify the most effective solutions to empower women, as well as to drive transformative change in current approaches to reduce IPV and promote gender equality in highly vulnerable populations in Colombia, and worldwide.

The goal of the project is to estimate the impact of generating livelihood opportunities and providing gender-based violence (GBV) training to reduce IPV among women in Colombia. This will generate much needed evidence on the most effective approach to empower women smallholder farmers and reduce their exposure to IPV. Investigators will conduct a cluster randomized controlled trial targeting approximately 100 smallholder farmers' associations and approximately 2700 women. Results will inform and strengthen future programming of humanitarian assistance and can be replicated in humanitarian interventions in other parts of the world.

The experimental operational research will compare two programmatic modalities and their impact on women's risk of exposure to IPV, against a comparison group where no intervention takes place. The modalities will include: (1) providing a stable income for women, and (2) providing a stable income and IPV trainings to women. The evaluation will take place in five departments: Cauca, Valle de Cauca, Meta, Caquetá, and Nariño.

ELIGIBILITY:
Inclusion Criteria:

* Women currently married or living together with a man as if married
* Males or females who are active within the farmer's association are eligible to participate

Exclusion Criteria:

* Women who have a husband/partner who is living elsewhere permanently

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1882 (Actual)
Dates: Start 2016-04-02 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence Physical and/or Sexual IPV | Post-Baseline (12 Months)
  The number of new physical and/or sexual IPV encounters as reported in the study survey.
Change in Prevalence of Physical and/or Sexual IPV | Baseline, End-Line (12 Months Post Intervention)
  The difference in the number of physical or sexual IPV encounters between baseline and post intervention as reported in the study survey.

SECONDARY OUTCOMES:
Incidence Physical IPV | Post-Baseline (12 Months)
  The number of new physical IPV encounters reported.
Incidence Sexual IPV | Post-Baseline (12 Months)
  The number of new sexual IPV encounters as reported in the study survey.
Incidence Psychological IPV | Post-Baseline (12 Months)
  The number of new physiological IPV encounters as reported in the study survey.
Incidence Economic Coercion | Post-Baseline (12 Months)
  The number of new encounters of economic coercion as reported in the study survey.
Change in Prevalence of Physical IPV | Baseline, End-Line (12 Months Post Intervention)
  The difference in the number of physical IPV encounters between baseline and post intervention as reported in the study survey.
Change in Prevalence of Sexual IPV | Baseline, End-Line (12 Months Post Intervention)
  The difference in the number of sexual IPV encounters between baseline and post intervention as reported in the study survey.
Change in Prevalence of Psychological IPV | Baseline, End-Line (12 Months Post Intervention)
  The difference in the number of psychological IPV encounters between baseline and post intervention as reported in the study survey.
Change in Prevalence of Economic Coercion | Baseline, End-Line (12 Months Post Intervention)
  The difference in the number of economic coercion encounters between baseline and post intervention as reported in the study survey.

OTHER OUTCOMES:
Women's Attitudes Towards Gender | End-Line (12 Months Post Intervention)
  General attitudes towards gender will be qualitatively collected via interview from women post intervention.
Change in Women's Economic Empowerment | Baseline, End-Line (12 Months Post Intervention)
  Changes in women's thoughts on economic empowerment will be qualitatively collected via interview.
Change in Women's Attitudes Towards Gender | Baseline, End-Line (12 Months Post Intervention)
  Differences in general attitudes towards gender will be qualitatively collected via interview from women from baseline to post intervention.
Household Food Insecurity | End-Line (12 Months Post Intervention)
  Access to adequate amounts of food for the household will be assessed via interview.
Change in Household Food Insecurity | Baseline, End-Line (12 Months Post Intervention)
  Change in access to adequate amounts of food for the household from baseline to end-line will be assessed via interview.
Total Personal and Household Income | End-Line (12 Months Post Intervention)
  The total income generated for a household will be collected via interview.
Change in Total Personal and Household Income | Baseline, End-Line (12 Months Post Intervention)
  The difference in the total income generated for a household from baseline to end-line.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Yount, PhD, Principal Investigator — Emory University
Locations (1):
- World Food Programme Colombia, Aurora, Bogota D.C., Colombia